CLINICAL TRIAL: NCT06647693
Title: Do Motor Synchrony Games Improve Self Regulation?
Acronym: MSG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Principal Investigator, George Wolford, Assistant Professor, Appalachian State University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HS-24-110
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Preschool Child; Executive Function (Cognition)
Keywords: Executive Function; Behavioral Self-Regulation; Autism; Preschool child
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Sequential is the best match for the intervention study model. The primary intervention model is a single case experimental design called a multiple baseline design. The investigators randomized participants into one of three start dates for the beginning of the intervention. Data is taken on a twice weekly basis during the baseline phase and intervention phase. The investigators also will add formal testing upon initial contact, right before intervention, upon completion of intervention procedures, and a follow-up without intervention.
Who Masked: Outcomes Assessor
Masking Description: Investigator and research assistant will not be blind. A second blinded research assistant will complete reliability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- First cohort (Experimental): These participants begin the intervention after 6 sessions
  Interventions: Behavioral: Motor Synchrony Games (MSG)
- Second cohort (Experimental): These participants enter the intervention after 9 baseline sessions
  Interventions: Behavioral: Motor Synchrony Games (MSG)
- Third cohort (Experimental): These participants enter the intervention after 12 baseline sessions (and 3 sessions post-hurricane Helene)
  Interventions: Behavioral: Motor Synchrony Games (MSG)

INTERVENTIONS:
Behavioral: Motor Synchrony Games (MSG) — The motor synchrony games (MSG) intervention uses fun but progressively more challenging gross motor and imitation games to promote behavioral self-regulation. Primary activities include: songs and fingerplays, stop and go games, and imitation games. These games get progressively more challenging over time by varying signal/modality. For example, going from a verbal and gestural paired "stop" and "go" signal to only a gestural stop signal. A fidelity checklist is used to ensure the intervention is appropriately used with the following criteria (uses >10 imitation trials, >10 Stop & Go games, >3 trials/min on average with >5 trials/min preferred, use of progressive challenge, opportunities for Child Choice, environmental arrangement, and therapeutic strategies such as modeling).

SUMMARY:
The goal of this study is to determine if progressively more challenging playground games (motor synchrony games) improve executive function in preschool-aged children.

DETAILED DESCRIPTION:
Self-regulation (SR) skills in early childhood predict later academic achievement and protect against developing internalizing and externalizing problems such as depressive symptoms or aggressive behavior (McClelland et al., 2019; Robson et al., 2020). One way to target SR skills is to use a program that involves motor synchrony games (e.g., musical freeze) (Gibb et al., 2021; McClelland et al., 2019; Zelazo et al., 2018). This study seeks to implement a similar motor synchrony games protocol in mixed ability groups to target SR. The investigators plan to use a multiple baseline design, a type of single case experimental design, to characterize the growth for individual participants.

The specific aims are as follows:

Aim 1: To determine if targeted motor synchrony games can achieve an increase in SR.

Aim 2: To examine how individual participants, including those with and without disabilities, respond to the protocol.

(Protocol modified in October:) Aim 3: Determine if hurricane Helene impacted the self-regulation of participants

Schedule: During the study, participants will begin baseline procedures twice a week for (approximately) 6, 9, 12 sessions (12 session group must have 3 sessions post-hurricane Helene). Afterwards, the participants will start the intervention. During baseline and intervention, the investigators measure their completion of a progressively more challenging stop and go task and imitations as the repeated measure. This procedure reflects a multiple baseline design.

As an exploratory analysis, all enrolled participants will complete assessments at 5 times: initial time point, before starting intervention, after hurricane Helene, after intervention procedures complete, and 2 months follow-up. (Post-hurricane data point was added due to the ~3 week shut down that disrupted the study in October. Parents could opt-out of these specific procedures.)

Intervention procedures: In the intervention period, participants will join the investigators in intervention sessions that last approximately 20-25 minutes and will involve rhythm and motor games or activities. All games are designed to have aspects of synchronous movement but should be fun and developmentally appropriate.

Following completion of the intervention, the investigators will graph the results for visual inspection of the stop and go and imitation data. The investigators also will calculate Tau-U statistics (including correcting for baseline trend).

The investigators plan to use the other assessment measures in two ways: the investigators will use an ANOVA to determine if there were significant differences between assessment time points. The investigators also will use a regression to account for the actual time that has passed.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the preschool classroom
* Express at least one word
* Runs independently

Exclusion Criteria:

* Known motor disorder
* Parents report the child cannot hear spoken language
* Parents report the child cannot see person gesturing 10 feet away

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Stop and Go Sequence | Twice weekly for approximately 12 weeks
  Participants are asked to "stop" and then "go" in progressively more challenging ways. The purpose is to measure self-regulation (specifically the inhibition executive function ability)
NIH Toolbox | Implemented 5 times - initial evaluation, before beginning intervention (~6, 9, or 12 sessions), post-hurricane Helene, approximately 12 weeks after initial evaluation, approximately 2 month follow-up)
  Card Sort & Picture Vocabulary. The purpose is to measure behavioral self-regulation / executive function (Card Sort) and also language (Picture Vocabulary)
Head, Toes, Knees, Shoulders - Revised | Implemented 5 times - initial evaluation, before beginning intervention (~6, 9, or 12 sessions), post-hurricane Helene, approximately 12 weeks after initial evaluation, approximately 2 month follow-up)
  HTKS-R (Gonzales, 2021). The purpose is to measure behavioral self-regulation.

SECONDARY OUTCOMES:
Imitation Score | Twice weekly for approximately 12 weeks
  Three trials of imitation. Scored as 2 - immediate and correct imitation, 1 - partial or delayed imitation, 0 - no imitation (for ~2 seconds). The purpose is to measure imitation/synchrony.
Patient reported outcome measures | Twice weekly for approximately 12 weeks
  Participants are asked each time if the intervention or baseline session was "fun," "not fun," "ok," or "sad". The purpose is to measure how the participants felt about the intervention and/or screen for unexpected results (e.g., all participants suddenly saying "sad" after a session)
BRIEF-P | Initial and about 12 weeks after (twice)
  Classroom teachers will complete the BRIEF-P. The purpose is to triangulate measurements of behavioral self-regulation / executive function
Stop latency | The investigators had initially planned four times (initial, after baseline, about 12 weeks after, and the two 2 month follow up), but due to mat availability, the investigators are only going to complete this outcome measure twice
  Using the Zeno Walkway system, the investigators will measure the latency in the participant's stops between when participants hear a beep signal and when participants stop

CONTACTS AND LOCATIONS:
Locations (1):
- Appalachian State University, Boone, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and outcome measures will be available on OSF ( https://osf.io/ ) following the completion of the study. The investigators plan to amend this record to add that link once present. Some data may be shared directly in a future manuscript.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within approximately a year after collection or pending publication.
Access Criteria: The data should be available on OSF and publicly available.